CLINICAL TRIAL: NCT05390489
Title: Effect of Arabica Coffee (Coffea Arabica) Cascara Pulp Extract From Gayo as Topical Antioxidant in the Treatment of Photoaging
Brief Title: The Effect of Arabica Gayo Cascara Pulp Extract on Photoaging
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wahyu Lestari (Other)
Responsible Party: Sponsor-Investigator, Wahyu Lestari, Assistant Professor, Universitas Syiah Kuala
Organization: Universitas Syiah Kuala (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 018/EA/FK-RSUDZA/2022
Record Dates: First submitted 2022-05-14; First posted 2022-05-25 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cascara pulp arabica gayo coffee cream (Experimental): The installation of a patch test for the cascara pulp cream of Gayo Arabica coffee with a concentration of 10% was carried out on the upper arm and waited for 30 minutes to see if there were any side effects. If no side effects occur, the patch test is left for 48 hours. After 48 hours, patch test was opened and the skin condition was assessed for irritation/redness and skin moisture. This condition was also re-evaluated at 72 and 96 hours later.
  Interventions: Drug: Cascara pulp arabica gayo coffee cream

INTERVENTIONS:
Drug: Cascara pulp arabica gayo coffee cream — extract of cascara pulp arabica gayo coffee

SUMMARY:
The purpose of this study was to assess the safety of Gayo Arabica coffee pulp extract cream as an antioxidant for the skin that can increase skin moisture

DETAILED DESCRIPTION:
This study is a phase I clinical trial aimed to assess the safety of the cream to be performed on volunteers, women, aged 20-40 years, who have healthy and normal skin. Research subjects that included in the study were determined based on inclusion and exclusion criteria. Enumerators previously provided information to the public using print media about this research to obtain research subjects that matched the inclusion and exclusion criteria. After that, the enumerators will conduct interviews and the willingness of research subjects according to the inclusion criteria by filling in the informed consent. Then before intervention, there will be an examination of skin conditions which will be carried out by two dermatologists including the condition of research subjects' skin moisture with a corneometer.

The cascara pulp cream of Gayo Arabica coffee works to improve skin structure and increase moisture in the skin. The safety test of the cream with the patch test method of cascara pulp cream of Gayo Arabica coffee was carried out by researchers and left for 48 hours. After 48 hours, the patch test unit was opened and evaluated by 2 dermatologists, the changes that occurred were recorded. Then with a corneometer examination was done to determine skin moisture. The same thing will also be done at the research subjects visit after 72 hours and 96 hours after the patch test is opened to reassess whether there are changes in the skin such as irritation/redness and skin moisture.

Data analysis in this study used univariate, bivariate and multivariate data analysis. Univariate analysis was carried out by describing the characteristics of the basic data in the form of frequency distribution, average value, standard deviation and range that occurred from the variables studied, both dependent (dependent) and independent (independent) variables. Bivariate analysis in this study was carried out by collecting data on a numerical scale first and then assessing its distribution using the Kolmogorov Smirnov test. Furthermore, if the data is normally distributed, the comparison of the mean before and after the intervention in the group will be analyzed using the Paired sample t-test. If the data is not normally distributed, a non-parametric test in the form of the Wilcoxon Rank test will be used.

ELIGIBILITY:
Inclusion Criteria:

* female, healthy and normal skin condition
* age 20-60 years old
* Willing to participate in research

Exclusion Criteria:

* history of allergy to one of the ingredient of the cream
* history of allergy to coffee

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
change in skin condition | 48 hours, 72 hours, 96 hours after patch test installation
  to observe any skin reaction to the cream using the International Contact Dermatitis Research Group (ICDRG) critera
change in Skin hydration | 48 hours, 72 hours, 96 hours after patch test installation
  skin hydration assessed by corneometer

CONTACTS AND LOCATIONS:
Overall Officials: Wahyu Lestari, Principal Investigator — wahyu_lestari2000@unsyiah.ac.id
Locations (1):
- dr. Zainoel Abidin General Hospital, Banda Aceh, Nanggore Aceh Darussalam, Indonesia

IPD SHARING:
Plan to Share IPD: No
to ensure the confidentiality of data obtained from respondents

REFERENCES:
- [Background] Quan T, Qin Z, Xia W, Shao Y, Voorhees JJ, Fisher GJ. Matrix-degrading metalloproteinases in photoaging. J Investig Dermatol Symp Proc. 2009 Aug;14(1):20-4. doi: 10.1038/jidsymp.2009.8. PMID 19675548
- [Background] Wasitaatmadja S. Pigmentasi Kulit FKUI, ed Dermatology Kosmetik. Published Online. 2011;7-12
- [Background] Chien AL, Qi J, Grandhi R, Kim N, Cesar SSA, Harris-Tryon T, Jang MS, Olowoyeye O, Kuhn D, Leung S, Rainer BM, Poon F, Suh J, Cheng N, Okoye GA, Kang S. Effect of Age, Gender, and Sun Exposure on Ethnic Skin Photoaging: Evidence Gathered Using a New Photonumeric Scale. J Natl Med Assoc. 2018 Apr;110(2):176-181. doi: 10.1016/j.jnma.2017.05.001. Epub 2017 Jun 7. PMID 29580452
- [Background] Iriondo-DeHond A, Elizondo AS, Iriondo-DeHond M, Rios MB, Mufari R, Mendiola JA, Ibanez E, Castillo MDD. Assessment of Healthy and Harmful Maillard Reaction Products in a Novel Coffee Cascara Beverage: Melanoidins and Acrylamide. Foods. 2020 May 12;9(5):620. doi: 10.3390/foods9050620. PMID 32408584
- [Background] Wen KC, Fan PC, Tsai SY, Shih IC, Chiang HM. Ixora parviflora Protects against UVB-Induced Photoaging by Inhibiting the Expression of MMPs, MAP Kinases, and COX-2 and by Promoting Type I Procollagen Synthesis. Evid Based Complement Alternat Med. 2012;2012:417346. doi: 10.1155/2012/417346. Epub 2011 Dec 1. PMID 22203872
- [Background] Andarina R, Djauhari T. Antioksidan dalam Dermatologi. J Kedokteran dan Kesehatan. 2017;4(1):39-48
- [Background] Thiele JJ. Oxidative targets in the stratum corneum. A new basis for antioxidative strategies. Skin Pharmacol Appl Skin Physiol. 2001;14 Suppl 1:87-91. doi: 10.1159/000056395. PMID 11509912
- [Background] Lestari W, Hasballah K, Listiawan MY, Sofia S. Identification of Antioxidant Components of Gayo Arabica Coffee Cascara Using the GC-MS Method. IOP Conference Series Earth Environmental Sciences. 2022;956(1):012011.
- [Background] Marcelinda A, Ridhay A. Aktivitas Antioksidan Ekstrak Limbah Kulit Ari Biji Kopi (Coffea sp) Berdasarkan Tingkat Kepolaran Pelarut The Atioxidant Activity Of Husk Coffea (Coffea sp) Extract Base On Various Levels Of Polar Solvent. Online J Nat Sci. 2016;5(1):21-30.
- [Background] Widiputri DI, Wijaya S, Kusumocahyo SP. Development of Skin Lotion Containing Antioxidant Extract from Coffee Pulp and Study on Its Stability. IOP Conf Ser Mater Sci Eng. 2020;742(1).
- [Background] Diamantina C. Utilization of Coffee Processing Waste in the Form of Antioxidant Skin Gel Containing Coffee Pulp Extract. 2015;15
- [Background] Yoon HS, Kim JR, Park GY, Kim JE, Lee DH, Lee KW, Chung JH. Cocoa Flavanol Supplementation Influences Skin Conditions of Photo-Aged Women: A 24-Week Double-Blind, Randomized, Controlled Trial. J Nutr. 2016 Jan;146(1):46-50. doi: 10.3945/jn.115.217711. Epub 2015 Nov 18. PMID 26581682
- [Background] Anggraeni Noviandini CRS. Patch Test dan Repeated Open Application Test ( ROAT ) pada Dermatitis Kontak Alergika ( Patch Test and Repeated Open Application Test ( ROAT ) in Allergic Contact Dermatitis ). Telaah Kepustakaan. 2014;220-8.